CLINICAL TRIAL: NCT01862965
Title: Treatment of Newly Diagnosed Moderate or Severe Chronic Graft-versus-host Disease With Prednisone and Everolimus (PredEver First) - A Prospective Multicenter Phase IIA Study -
Brief Title: Treatment of Newly Diagnosed Moderate or Severe Chronic Graft-versus-host Disease With Prednisone and Everolimus
Acronym: PredEver first
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Novartis (Industry); Crolll Gmbh (Other)
Responsible Party: Principal Investigator, PD Dr. med. Francis Ayuketang Ayuk, PD Dr. med., Universitätsklinikum Hamburg-Eppendorf
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PredEver first; 2011-004847-35 (EudraCT Number)
Record Dates: First submitted 2013-05-01; First posted 2013-05-27 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Chronic Graft-versus-host Disease
Keywords: firstline; treatment; prednisone; everolimus
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PredEver (Experimental): Prednisone and Everolimus
  Interventions: Drug: PredEver

INTERVENTIONS:
Drug: PredEver — Firstline treatment with prednisone and Everolimus

SUMMARY:
In this study patients with moderate to severe chronic graft-versus-host disease will be treated with a combination of prednisone and everolimus. Patients will be treated on the study for a maximum of 12 months and followed up for another 12 months.

The primary hypothesis of this study is that the addition of everolimus to prednisone increases response rates without increasing treatment related mortality or mortality due to relapse of underlying disease.

DETAILED DESCRIPTION:
Background

2.1 Chronic graft-versus-host disease

Chronic graft-versus-host disease (cGvHD) is the most common long-term complication of allogeneic hematopoietic stem cell transplantation (allo-HSCT), with an incidence of up to 70% in recipients of peripheral blood stem cells. Chronic GvHD is associated with impaired immunity, compromised functional status and quality of life and is besides relapse of underlying malignancy still the leading cause of morbidity and mortality beyond day 100 after allo-HSCT. The pathophysiology of cGvHD is still not well understood, however efforts made in the last years indicate a role of persistent allo-reactive T cells, B cells that produce auto- or allo-antibodies against the host antigens as well as donor antigen presenting cells (APC) that replace host APCs thus leading to indirect antigen presentation of allo-antigens. Persistent alloreactivity may be due to defective peripheral and central tolerance mechanisms as a result of failure of control by regulatory T cells (Tregs) and/or impaired negative selection of T cells in the thymus.

Corticosteroids have constituted the backbone of treatment of cGvHD over the past 4 decades. Addition of calcineurin inhibitors (CNI) to steroids in first-line therapy did not lead to significant improvement of response or patient outcome. The expanding therapeutic arsenal of cGvHD also includes many other agents which have been evaluated in second-line therapy such as mTOR inhibitors, extracorporeal photopheresis, mycophenolate mofetil, rituximab, alemtuzumab, thalidomide, imatinib, pentostatin, low dose methotrexate amongst others. The median duration of immunosuppression of 23 months and the high 3 year non-relapse mortality of up to 40% emphasize the urgent need for new first line treatment strategies.

3 Study rationale

The outcome of patients with chronic GvHDcGvHD treated with corticosteroids alone or in combination with CNI like CSA or tacrolimus is still very unsatisfactory with an increased relative risk of non-relapse mortality of up to 7 times compared to patients without or only mild cGvHD. While corticosteroids are generally accepted to be the backbone of systemic therapy, the role of CNI remains questionable. There is thus urgent need for improvement of first-line treatment of these patients. mTOR inhibitors like sirolimus (rapamycin) or everolimus have been shown to be effective in second-line treatment of cGvHD. In the light of these data and given the unmet medical need in the treatment of cGvHD, there is a rationale to examine the efficacy of an mTOR inhibitor in first line treatment of these patients with cGvHD.

4 Hypothesis and study objectives

The primary hypothesis of this study is that the addition of everolimus to prednisone increases response rates without increase ofincreasing non-relapse and relapse mortality. In contrast to CNI, everolimus may also facilitate the development of tolerance and thereby improve the durability of response, thus increasing the time to treatment failure.

4.1 General objectives

The main objective of this study is to investigate the clinical benefit of treatment with prednisone and everolimus in patients with chronic GvHDcGvHD. Treatment change or time to flare-up of cGvHD symptoms has been shown to correlate with survival of patients with cGvHD. In this study the addition of secondary treatment will reflect treatment failure and serve as a parameter for measuring clinical benefit.

6.3 Discussion of study design

Chronic GvHD occurs in about 50% of patients after allogeneic HSCT, more than 80% of whom will have moderate or severe disease requiring systemic therapy. The participation of 6 centres enables the recruitment of 60 patients within 24 months. The follow-up period of 1 year is sufficient to evaluate time to progression, which has been shown to predict survival. There is no control group. The findings of this study will be analysed and discussed in the light of historical data and lay the groundwork for a possible randomized study.

The German-Swiss-Austrian GvHD-group will run a registry prospectively documenting cGvHD cases, their treatment and outcome as from 2012. The control population will consist of patients treated in the cGvHD registry within the same time period as in this study. A comparison to the historical population treated in the placebo arm of the impact of Myfortic® in first line treatment of cGvHD [Martin et al.,2009] will also be performed.

7.4 Sample size estimation

The sample size estimation is based on data from the placebo arm of the randomized trial led by Paul Martin evaluating the impact of additional MMF in the initial treatment of cGvHD [data kindly provided by Paul Martin].

The rate of treatment success at 6 months in the placebo arm of the study (standard treatment with prednisone alone or prednisone plus a calcineurin inhibitor) was 62%.

Assuming a treatment success rate of 65% for patients receiving standard therapy (steroids alone or steroids and calcineurin inhibitor) and testing whether the combination of prednisone and everolimus would improve the rate of treatment success to 85%, with 80% power and a one-sided type error (α) of 5%, then at least 57 patients will need to be recruited. This study thus plans to recruit a total of 60 patients. This patient number will enable both comparison with patients treated during the same period within the planed cGvHD registry as well as a historic comparison with data from the above mentioned study led by Paul Martin.

8 Diagnosis and grading of cGvHD

8.1 Overview

Diagnosis and grading of cGvHD will be according to NIH consensus-criteria. If diagnosis of cGvHD depends on skin manifestations, an assessment of a biopsy should be organized by each site itself according to local routine. A central review is recommended but not obligatory.

8.2 Definition of high-risk cGvHD

High risk cGvHD is defined by one or more of the following criteria being fulfilled at time of diagnosis of cGvHD:

* < 100,000/µl platelets
* progressive onset of cGvHD (see 7.2.1 for definition)
* involvement of > 50% of total body surface area
* bilirubin > 2 mg/dl
* bronchiolitis obliterans

8.2.1 Definition of progressive onset cGvHD

Progressive onset cGvHD is defined as acute GvHD preceding cGvHD whereby either

1. no complete response (CR) of acute GvHD is attained before onset of cGvHD or
2. the time between CR of aGvHD and onset of symptoms of cGvHD is less than 2 weeks.

9.3 GvHD prophylaxis and acute GvHD therapy

9.3.1 GvHD prophylaxis

Any kind of GvHD prophylaxis may have been used, including mTOR-containing regimens. Type of GvHD prophylaxis will be documented and included in the analysis.

9.3.2 Acute GvHD therapy

Any kind of acute GvHD therapy may have been used, excluding mTOR inhibitors (everolimus or sirolimus).

9.3.3 Conditioning regimen and stem cell source

* Any kind of conditioning regimen (myeloablative or reduced intensity) may have been used for transplantation
* Stem cell source may have been bone marrow, peripheral blood stem cells or cord blood
* Donors may have been related or unrelated, matched or mismatched Conditioning intensity, stem cell source donor type and donor/recipient histocompatibility will be documented and included in analysis.

9.6 Patients' evaluation

9.6.1 Assessment of pre-registration characteristics

Prior to enrolment in the study patients will be examined for inclusion and exclusion criteria. A comprehensive assessment of organ involvement shall be performed according to the NIH consensus criteria. The time between this examination and the initiation of study treatment should be maximum 14 days.

9.7 Study monitoring

9.7.1 Clinical assessment visits

Regular clinical assessment visits are planned to include patient's physical examination, blood counts, blood chemistry and everolimus level.

9.7.2 Response assessment visits

Response to treatment will be assessed after 2 weeks, month 1, 3, 6, 9, and 12 after initiation of treatment, before introduction of secondary treatment and in case of premature study withdrawal. Response assessment will be performed prospectively as described in the publication by Martin et al. and retrospectively according to NIH consensus recommendations.

9.7.3 End of study assessment visits

Patients going off protocol regularly (after complete response or max. 1 year of treatment) or prematurely will undergo response assessment as outlined in section 8.7.2.

11 Treatment plan

11.1 Overview

After diagnosis of cGvHD patients will receive prednisone 1 mg/kg BW orally and everolimus (whole tablets or dispersible tablets) orally (targeted trough level 3-8 µg/l). Prednisone may also be administered intravenously at 1 mg/kg if patients are unable to take the oral formulation. Patients will be treated on the protocol for a maximum of 12 months. Patients still responding can continue with treatment off protocol at the discretion of the local physician. Patients will be followed-up for another 12 months after their end of protocol treatment.

11.2 Regular dosing and tapering of immunosuppressive drugs

11.2.1 Stopping of prior calcineurin inhibitors

If the patient is on a calcineurin inhibitor at time of study inclusion, CNI should be tapered and stopped within 1-3 weeks of initiation of study treatment, with an initial reduction of 50% at initiation of everolimus. The CNI baseline level should be not higher than 100 µg/ml for CSA and not higher than 6 µg/ml for tacrolimus after start of everolimus.

11.2.2 Stopping of prior mTOR inhibitors

If the patient is on sirolimus or everolimus prophylaxis at time of study inclusion, everolimus will be continued; sirolimus will be switched to everolimus without tapering or loading.

11.2.3 Dosing and recommended tapering of steroids

The initial dose of prednisone is 1 mg/kg BW given as a single dose in the morning. It is recommended to maintain this dose for at least 2 weeks and then taper depending on the patient's response (CR or PR), according to appendix 13.1 and 13.2. These tapering recommendations are meant to guide tapering speed. Patients with progressive disease after 2 weeks (> 25% in any organ) will be considered steroid-refractory and require secondary therapy.

11.2.4 Dosing and tapering of everolimus

The initial dose of everolimus will be 0.75 mg twice daily. The dose shall be adjusted to a targeted trough serum level of 3-8 µg/l, measured by HPLC or immunoassay 4 to 5 days after the previous dose change. Initial dose reduction may be considered in the presence of a co-medication interfering with metabolism of everolimus (see also 10.3.7.) Dose adjustments shall be according to clinical judgement of the local physician taking into consideration toxicity, serum levels and concomitant medication. Since CNI (particularly CSA) interact with everolimus, trough levels of everolimus will need to be readjusted after stopping CNI.

In patients with abnormal liver function tests the initial dose of everolimus will be 0.25 mg twice daily (see Appendix 13.5.5). Increment of daily dose should not surpass 0.5 mg within 1 week and initial monitoring of everolimus levels should be twice weekly until stable levels are attained for 2 weeks. This close monitoring will be repeated in case of any further dose modification. In patients who develop abnormal liver functions (as above) while already under treatment with everolimus, serum levels of the drug also need to be monitored closely (twice weekly), for at least 2 weeks after emergence of abnormal liver function to enable prompt dose modification if required.

After discontinuation of prednisone, patients should be monitored for at least 4 weeks for possible recurrence of cGvHD symptoms. In the absence of cGvHD activity, everolimus will be tapered off over a period of 12 to 24 weeks at the discretion of the local physician.

11.2.5 Concomitant therapy

Additional treatment with topical immunosuppressants like steroids is not considered treatment failure and can be given at the discretion of the local physician. Addition of secondary systemic immunosuppressive therapy is considered treatment failure as outlined in 4.1. Prophylaxis of infections, red blood cell and platelet support and antithrombotic prophylaxis will be given according to institutional practice. Monitoring for cytomegalovirus reactivation and preemptive therapy with antiviral agents will be performed according to centres' policy.

Documentation of adverse events and concomitant medications for each patient will be performed from the time a patient signs the informed consent form until the patient completes, withdraws or is withdrawn from the study.

11.3 Management of toxicity and dose modifications

11.3.1 Toxicity evaluation

Toxicity will be monitored at least once every month. Monitoring will include physical examination, laboratory liver and kidney function tests, blood lipids and blood counts.

11.3.2 Management of hyperlipidaemia

Patients with hyperlipidemia should be advised to maintain a diet. They should also receive HMG-CoA reductase inhibitors or fibrates. However caution must be taken and patients monitored for development of rhabdomyolysis. Everolimus should be continued during the treatment of hyperlipidaemia unless the lipid levels are uncontrollable with standard therapy. Dose modifications of everolimus for hyperlipidaemia and after diet and appropriate treatment with HMG-CoA reductase inhibitors or fibrates should be according to appendix 13.5.3

11.3.3 Management of TMA

TMA shall be documented and reported immediately. In the event of TMA, everolimus shall be discontinued. Plasmapheresis may be used at the discretion of the managing physician. Prevention of TMA involves avoiding drug levels above target range. High drug levels should prompt closer monitoring of hematocrit, platelets, LDH, BUN, creatinine and schistocytes.

11.3.4 Management of hematotoxicity

Patients with severe cGvHD often have cytopenia. Cytopenia may also be caused by concomitant medication like antiviral drugs or antibiotics or cGvHD itself. Dose modification of everolimus will therefore take baseline platelet counts into consideration. Absolute neutrophile count (ANC), hematocrit and platelet counts shall be monitored regularly. If other causes of cytopenia have been ruled out, everolimus dose will be modified according to appendix 13.5.4. GCSF, blood and platelet transfusions may be given at discretion of the local physician.

11.3.5 Management of non-infectious pneumonitis (NIP)

Symptoms of NIP usually subside completely within one month after cessation of treatment. This reversibility will enable differentiation from BOOP. The incidence and outcome of NIP will be documented and assessed in this study. Treatment with everolimus will not be restarted after diagnosis of NIP.

11.3.6 Management of other toxicities

Patients will also be monitored for other toxicities such as edema, arthralgias or aphthous ulcers. Efforts will be made to rule out other causes. If other causes of toxicity have been ruled out and toxicity is thought to be caused by everolimus and is significant, everolimus dose will be decreased to 50%. If symptoms do not improve or resolve after 2 weeks, everolimus will be held. If symptoms improve or resolve, everolimus will be restarted at 50% and gradually increased to full dose as tolerated. Everolimus can be held for a maximum of 14 successive days with the patient remaining on study, longer treatment breaks will mean premature termination of study treatment.

11.3.7 Other important considerations

Serum levels of everolimus are significantly influenced by food intake, thus everolimus should be taken at consistent times of the day consistently with or without food to minimize variability.

In appendix 13.5.1 and 13.5.2 drugs are listed which are known to interact with everolimus and/or prednisone. During concomitant medication with these drugs, caution should be taken and patients seen, at least once weekly to once every two weeks in order to closely monitor drug levels and perform clinical examinations for toxicity. Concomitant treatment not recommended should only be administered if deemed absolutely necessary.

Grapefruit juice or St. John's Wort must not be taken during treatment with everolimus.

Concomitant treatment with voriconazole is not recommended and should be avoided. If use of voriconazole is deemed absolutely clinically necessary, dose reduction of everolimus of up to 90% may be necessary. Concomitant treatment with other azoles like fluconazole or posaconazole also requires caution including closer monitoring of everolimus serum levels and dose adjustments. Concomitant treatment with atorvastatin, pravastatin or other HMG-CoA reductase inhibitors or fibrates requires monitoring of patients for signs of rhabdomyolysis and everolimus levels. Patients receiving Ciclosporin or tacrolimus will have these tapered and stopped as described in chapter 10.2.1. Everolimus dose will be adjusted thereafter according to serum levels.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's written informed consent
2. Women and men capable of reproduction must agree to use adequate contraceptive measures (condom, intrauterine devices, oral contraceptives) until three months after termination of treatment
3. Age ≥ 18 years
4. Diagnosis of classic chronic GvHDcGvHD according to NIH criteria [33] and fulfilment of criteria for moderate or severe cGvHD or o Diagnosis of overlap syndrome according to NIH criteria [33] and fulfilment of criteria for moderate or severe cGvHD and ≤ clinical grade 2 of acute GvHD of the gut and no grade 4 acute GvHD of the skin.

NB: A maximum of 30 patients with overlap syndrome will be included in the trial.

Exclusion Criteria:

1. Late persistent or recurrent acute GvHD without evidence of cGvHD
2. Relapsed or progressive malignant disease (other than minimal residual disease diagnosed by molecular methods)
3. Severe uncontrolled infections
4. Pregnant or lactating women
5. Inability to tolerate 1 mg/kg prednisone
6. Inability to take oral medication
7. Known hypersensitivity to everolimus
8. History of mTOR- inhibitor associated non-infectious pneumonitis
9. Participation in another interventional clinical trial with intervention within < 30 days
10. Prior use of mTOR- inhibitor (everolimus or sirolimus) for treatment of acute GvHD
11. Prior systemic treatment for chronic GvHD>of cGvHD ≥ 72h
12. Psychiatric illness that would prevent granting of informed consent
13. Active viral infection with HIV, hepatitis B or hepatitis C
14. Severe cardiovascular disease (uncontrolled arrhythmias, congestive heart failure NYHA III or IV, or symptomatic ischemic heart disease)
15. History of mTOR- inhibitor or CNI-associated TMA that led to discontinuation of mTOR- inhibitor or CNI
16. Patients with neutrophils < 1000 1,000/µl and / /or platelets < 20.,000/ul µl at time of screening
17. Donor lymphocyte infusion within the last 30 days
18. Pre-existing hyperlipidemia prior to treatment with calcineurin inhibitor or mTOR inhibitor
19. Wound healing complications
20. Active lymphoma as well as other malignancies
21. Edema (angioneurotic or peripheral)
22. Peptic ulcer
23. Severe colitis ulcerosa
24. Diverticulitis
25. Severe osteoporosis
26. Poorly- controlled hypertension
27. Glaucoma (angle closure or open angle)
28. Cornea ulcer or cornea-injuries
29. Severe diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-03-06 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
rate of treatment success | at 6 months
  Patient being alive and having achieved a CR or PR of cGvHD without addition of secondary systemic treatment for cGvHD (see below) and without development of relapse of underlying disease. Addition of any immunosuppressive or immunomodulatory systemic therapy aimed at treating or controlling symptoms of chronic GvHDcGvHD is considered treatment failure. Examples of secondary systemic therapies include (but are not limited to) cyclosporine ACSA, tacrolimus, methotrexate, mycophenolate, rituximab, azathioprine, pentostatine, cyclophosphamid, chloroquine, imatinib, dasatinib, thalidomide, alemtuzumab, etanercept, antithymocyte globulin, infliximab, basiliximab, daclizumab, extracorporeal photopheresis, psoralen with UVA-irradiation (PUVA), pulsed steroid exceeding a dose of 2 mg/kg/day.

SECONDARY OUTCOMES:
the overall survival rate of patients treated with prednisone and everolimus for chronic GvHDcGvHD | 1 year
time to treatment failure | average time up to 12 months from start of treatment
  To evaluate the time to treatment failure, treatment failure being defined as progression of cGvHD after ≥ 2 weeks in any organ, lack of response (CR/PR) after 12 weeks and/or addition of secondary systemic treatment for cGvHD.
speed of response | average time up to 12 months from start of treatment
  To evaluate the speed of response (time to achievement of CR or PR) of patients treated with prednisone and everolimus for chronic GvHD
Relapse of underlying disease | 1 year
  To evaluate the relapse rate of underlying malignancies of patients treated with prednisone and everolimus
side effects | 1 year
  To assess the side effects of prednisone and everolimus in patients with cGVHD

OTHER OUTCOMES:
Safety endpoints | 1 year
  All adverse events shall be documented and assessed in this study as described in section 9 below. Particular emphasis will be made on the following:
  * Thrombotic microangiopathy (TMA)
  * Non-infectious pneumonitis (NIP)
  * Avascular osteonecrosis

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Jena, Jena
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Klinikum der Universität Regensburg, Regensburg
  - Universitätsklinikum Ulm, Ulm
  - Deutsche Klinik fuer Diagnostik GmbH, Wiesbaden